CLINICAL TRIAL: NCT07236944
Title: Pivmecillinam as Oral Step-Down Treatment for Escherichia Coli Febrile Urinary Tract Infection Versus Standard of Care: A Randomized Controlled Non-Inferiority Multicenter Trial
Brief Title: Pivmecillinam as Oral Step-Down Treatment for Escherichia Coli Febrile Urinary Tract Infection Versus Standard of Care
Acronym: PIVOT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: The Swedish Research Council (Other Government); Uppsala Clinical Research Center, Sweden (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PIVOT; 2023-503447-33-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Febrile Urinary Tract Infection
Keywords: Urinary Tract Infection; Pivmecillinam; Escherichia coli
MeSH Terms: conditions — Urinary Tract Infections; Escherichia coli Infections | interventions — Amdinocillin Pivoxil; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (Active Comparator): The control group will receive standard of care treatment at the discretion of the responsible physician and according to existing treatment guidelines.
  Interventions: Drug: Standard of Care (Investigator Choice)
- Pivmecillinam (Experimental): Pivmecillinam (high dose, 400 mg four times daily).
  Interventions: Drug: Pivmecillinam

INTERVENTIONS:
Drug: Pivmecillinam — Patients randomized to pivmecillinam will be provided with 400 mg tablets for 3 to 8 days of treatment, to be taken four times daily, resulting in a total treatment duration of 7 or 10 days (including the initial 2-4 days of intravenous treatment). The shorter treatment duration of 7 days will be used for female patients with no complicating factors (structural or functional urologic abnormalities, urinary tract catheterization, and diabetes mellitus). The longer treatment duration of 10 days will be used for all other patients.
  Arms: Pivmecillinam
Drug: Standard of Care (Investigator Choice) — The control group will receive standard of care antibiotic treatment at the discretion of the responsible physician and according to existing treatment guidelines, with a total treatment duration of 7 to 14 days. The following antibiotics will be considered adequate. Intravenous antibiotics: 1) Penicillins; ampicillin, piperacillin/tazobactam, 2) cephalosporins; cefotaxime, cefuroxime, ceftriaxone, 3) carbapenems; ertapenem, imipenem, meropenem, 4) monobactams; aztreonam, 5) aminoglycosides; amikacin, gentamicin, tobramycin, 6) other; fosfomycin. Oral antibiotics: 1) ciprofloxacin, 2) trimethoprim-sulfamethoxazole, 3) amoxicillin or amoxicillin/clavulanic acid provided that the isolated E. coli is determined susceptible according to the EUCAST-breakpoint for systemic infections, i.e., MIC ≤ 8 mg/l, and high dosing is used (≥750 mg amoxicillin x 3 and ≥750 mg amoxicillin/125 mg clavulanic acid x 3, respectively) and 4) tebipenem (if approved by the EMA).
  Arms: Standard of care

SUMMARY:
The goal of this clinical trial is to learn if oral treatment with pivmecillinam is effective to treat febrile urinary tract infections in adult patients. Hospitalized patients who have received 2-4 days of intravenous antibiotic therapy for febrile urinary tract infections, and have responded to treatment, will be randomized to either pivmecillinam or standard treatment (other oral or intravenous antibiotics).

The main question the study aims to answer is if oral follow-up with pivmecillinam is as effective as standard treatment. Patients will be evaluated for clinical response (resolution of fever and urinary tract symptoms) and microbiological response (no growth of bacteria in urine) 7 and 28 days after the end of treatment. Patients will also be asked about side effects. Some of the participants will also be examined for changes in the gut microbiome and drug exposures in blood and urine.

Participants will:

1. Keep a patient diary to record antibiotic intake, body temperature, urinary tract symptoms, and suspected side effects until 7 days after end of treatment.
2. Participate in phone interviews 7 and 28 days after end of treatment to assess clinical response.
3. Provide urine samples 7 and 28 days after end of treatment to evaluate microbiological response.
4. A subgroup (60 patients) will provide fecal samples at five time-points over three months to assess antibiotic-induced changes in the gut microbiome.
5. A subgroup (30 patients) treated with to pivmecillinam will provide blood and urine samples to determine the pharmacokinetics of mecillinam during one dosing interval.

DETAILED DESCRIPTION:
Background:

Escherichia coli is the predominant uropathogen and the most common cause of bloodstream infections. In the hospital setting, patients with febrile UTI (fUTI) are normally treated with intravenous antibiotics for 2-4 days until clinical improvement followed by oral step-down treatment guided by microbiological antibiotic susceptibility testing results. However, oral treatment options are increasingly limited due to emerging resistance in uropathogens and the lack of new antibiotics.

This non-inferiority, open label, randomized clinical trial (RCT), conducted in Sweden and Norway, will evaluate the efficacy of an oral narrow-spectrum penicillin (pivmecillinam) as oral step-down for patients with fUTI caused by Escherichia coli. Pivmecillinam is a first line antibiotic for acute cystitis and is sometimes used also for fUTI in Denmark and Norway although no previous RCT has evaluated its efficacy for this indication. Pivmecillinam will be compared to standard of care, i.e. step-down treatment with other orally administered antibiotics, such as ciprofloxacin or trimethoprim-sulfamethoxazole, or continued intravenous antibiotic treatment. The target sample size is 560 participants, to be enrolled over a three-year period.

Patient population:

The following PICO (Population/Intervention/Control/Outcome) applies: Population - Patients with E. coli fUTI receiving initial intravenous antibiotic treatment; Intervention - Oral follow-up treatment with pivmecillinam; Control - Standard of care; Outcome - Clinical response (primary endpoint).

Objectives:

The primary objective is to investigate if the clinical response with oral follow-up treatment with pivmecillinam 400 mg four times a day (QID) is non-inferior to standard of care in patients with E. coli fUTI 7 (+/-2) days after end of treatment (EOT).

Secondary objectives are to investigate treatment effects on:

1. Sustained clinical response 28 days after EOT
2. Microbiological response 7 days after EOT
3. Sustained microbiological response 28 days after EOT
4. Adverse events up to 7 days after EOT
5. Disturbances in the intestinal microbiome (60 patients) up to 3 months after EOT
6. Pharmacokinetics of mecillinam in plasma and urine (30 patients) during one dosing interval
7. Cost effectiveness of pivmecillinam compared to standard treatment

Primary endpoint:

The primary endpoint is defined as clinical response, defined as: i) no new healthcare contacts or antibiotic treatments for suspected or proven UTI, ii) sustained defervescence (< 38°C), and iii) patient-documented resolution of fUTI symptoms that were present and recorded in the eCRF at trial entry (and no new fUTI symptoms) at test of cure (TOC), which will be performed 7 (+/-2) days after EOT. The evaluation of clinical response (primary endpoint) will be performed by blinded assessors.

Statistical analysis:

Non-inferiority will be defined as < 10% lower clinical response at TOC. The primary analysis will be based on all randomized patients (intention-to-treat, ITT). Per-protocol (PP) analysis will be performed as supplementary analysis, and the consistency of ITT and PP results will be evaluated. Assuming 80% clinical response rate in both arms, a non-inferiority limit of 10%-points, 1:1 randomization, and 10% loss to follow-up, 280 patients in each arm (total 560 randomized patients) would give 80% power to detect non-inferiority at a one-sided alpha=0.025.

Intervention and control group:

Patients with fUTI caused by E. coli treated with adequate intravenous antibiotics for 2-4 days will be randomized to i) oral step-down treatment with pivmecillinam (high dose, 400 mg QID), or ii) standard of care. Patients randomized to pivmecillinam will be provided with tablets for a total treatment duration of 7 (female patients with no complicating factors) or 10 days (all other patients).

The control group will receive standard treatment, as determined by the responsible physician in accordance with current treatment guidelines and guided by the antibiotic susceptibility testing results of the isolated pathogen. The total treatment duration will be 7 to 14 days. In Norway, where pivmecillinam is already recommended for some patients with fUTI, participants randomized to the control group can be prescribed any antibiotic considered standard of care except for pivmecillinam. The following antibiotics will be considered adequate if the isolated bacteria are reported susceptible to the prescribed drug by the clinical microbiological laboratory. Intravenous antibiotics: 1) Penicillins; ampicillin, piperacillin/tazobactam, 2) cephalosporins; cefotaxime, cefuroxime, ceftriaxone, 3) carbapenems; ertapenem, imipenem, meropenem, 4) monobactams; aztreonam, 5) aminoglycosides; amikacin, gentamicin, tobramycin, 6) other; fosfomycin. Oral antibiotics: 1) ciprofloxacin, 2) trimethoprim-sulfamethoxazole, 3) amoxicillin or amoxicillin/clavulanic acid provided that the isolated E. coli is determined susceptible according to the EUCAST breakpoint for systemic infections, i.e., MIC ≤ 8 mg/l, and high dosing is used (≥750 mg amoxicillin x 3 and ≥750 mg amoxicillin/125 mg clavulanic acid x 3, respectively) and 4) tebipenem (if approved by the EMA).

Diagnostic and monitoring procedures:

TOC will be performed 7 (+/- 2) days after EOT by phone interview. A second follow-up will be performed 28 (+/- 2) days after EOT to assess sustainable clinical response. Urine samples will be collected 7 and 28 days after EOT to evaluate microbiological response.

Fecal samples for microbiome analysis will be collected from 30 patients treated with pivmecillinam and 30 patients treated with ciprofloxacin at the time of randomization (prior to oral treatment), at EOT, and 7 days, 28 days, and 3 months after EOT (±2 days).

The pharmacokinetics of mecillinam in plasma and urine will be assessed in 30 patients treated with pivmecillinam. Blood samples will be drawn in conjunction with the third dose or later, at 0 h (before dose), and 1 h, 2 h, 4 h and 6 h (after dose). Urine sampling will be performed within one dosing interval after ≥3 doses during 0-3 h and 3-6 h.

Risk/benefit assessment:

Pivmecillinam is commonly used and proven safe for uncomplicated cystitis, and the risks of study participants is considered very low. If pivmecillinam shows non-inferiority to standard of care, the results of the study will benefit patients with fUTI as well as health care and society at large. A shift to oral treatment means shorter hospitalization and no need for repeated visits or intravenous catheters, thereby reducing suffering, the risk of healthcare-associated infections, and costs. Using a narrow-spectrum antibiotic instead of broad-spectrum antibiotics reduces the risks of side effects and emergence and spread of resistant bacteria. The study will also provide a better understanding of the relative collateral damage of the study drugs on the microbiome and pivmecillinam pharmacokinetics, which will inform future treatment decisions and dosing.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age.
2. Diagnosis of fUTI, defined as i) fever ≥ 38°C and ii) at least one of the following: flank pain or pelvic pain, nausea or vomiting, dysuria, urinary frequency or urgency, and costovertebral angle tenderness on physical examination.
3. Growth of E. coli in urine with antimicrobial susceptibility to mecillinam.
4. Adequate intravenous antibiotic treatment for fUTI (defined below) for 2 days to which the isolated E. coli is determined susceptible.
5. Defervescence and hemodynamic stability for at least 24 hours, according to the responsible physician.
6. Planned treatment with one of the following antibiotics, should the patient be randomized to the standard-of-care arm. Intravenous antibiotics: 1) Penicillins; ampicillin, piperacillin/tazobactam, ≥2) cephalosporins; cefotaxime, cefuroxime, ceftriaxone, 3) carbapenems; ertapenem, imipenem, meropenem, 4) monobactams; aztreonam, 5) aminoglycosides; amikacin, gentamicin, tobramycin, 6) other; fosfomycin. Oral antibiotics: 1) ciprofloxacin, 2) trimethoprim-sulfamethoxazole, 3) amoxicillin or amoxicillin/clavulanic acid provided that the isolated E. coli is determined susceptible according to the EUCAST-breakpoint for systemic infections, i.e., MIC ≤ 8 mg/l, and high dosing is used (≥750 mg amoxicillin x 3 and ≥750 mg amoxicillin/125 mg clavulanic acid x 3, respectively) and 4) tebipenem (if approved by the EMA).
7. Signed informed consent.

Exclusion Criteria:

1. Adequate intravenous antibiotic treatment for > 4 days prior to randomization or other adequate (microbiologically active) oral antibiotic treatment for the same fUTI episode prior to recruitment.
2. Growth of other bacterial species than E. coli, or fungi, in urine.
3. Contraindication for pivmecillinam (e.g. allergy).
4. Clinical suspicion of bacterial prostatitis.
5. Renal abscess.
6. Kidney transplant.
7. Myelosuppressive disorder with neutrophil count < 0.5 x 10(9)/L at randomization.
8. Planned antibiotic treatment for fUTI > 14 days.
9. Likely to be prescribed antibiotic prophylaxis after treatment.
10. Other intravenous or oral antibiotic treatment; ongoing or planned during the follow-up period (i.e. until 28 days after EOT for fUTI).
11. Severe renal impairment (eGFR < 20 mL/min) at randomization.
12. Morbid obesity (BMI > 40 kg/m2).
13. Pregnancy or breastfeeding.
14. Unlikely to follow instructions or the study protocol.
15. Previous participation in the study.
16. If consenting to microbiome analysis: i) contraindication for ciprofloxacin (e.g. allergy), ii) unlikely to be able to provide fecal samples per protocol, iii) treatment with antibiotics in the past 3 months before the current fUTI episode, iv) chronic intestinal disease or previous surgery in the gastrointestinal tract.
17. If consenting to pharmacokinetic analysis: expected difficulties in providing blood and urine samples per protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Clinical response (primary endpoint). | 7 (+/-2) days after EOT
  Clinical response: i) no new healthcare contacts or antibiotic treatments for suspected or proven UTI, ii) sustained defervescence (< 38°C), and iii) patient-documented resolution of fUTI symptoms that were present and recorded in the eCRF at trial entry (and no new fUTI symptoms) at test of cure (TOC), which will be performed 7 (+/-2) days after end of treatment (EOT).
  The evaluation of clinical response (primary endpoint) will be performed by blinded assessors.

SECONDARY OUTCOMES:
Sustained clinical response | 28 (+/- 2) days after EOT
  Sustained clinical response: i) no new healthcare contacts or antibiotic treatments for suspected or proven UTI, ii) no recurrent fever (≥ 38°C), and iii) no recurrent UTI symptoms after completion of the initial therapy and until 28 (+/- 2) days after EOT.
Microbiological response | 7 (+/-2) days after EOT
  Microbiological response: no detectable growth of E. coli in urine sampled at TOC, i.e., 7 (+/-2) days after EOT.
Sustained microbiological response | 28 (+/- 2) days after EOT
  Sustained microbiological response: no detectable growth of E. coli in urine sampled at the second follow-up 28 (+/- 2) days after EOT.
Occurrence and severity of adverse events | From start of study treatment until test of cure 7 (+/-2) days after EOT
  Occurrence and severity of adverse events from start of study treatment until TOC; recorded by the participants in a study diary, documented in the medical records, or reported at the TOC follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Tängdén, MD, Professor, Principal Investigator — Department of Medical Sciences, Uppsala University
Locations (13):
- Norway (2):
  - Haukeland University Hospital, Haukeland
  - Oslo University Hospital, Oslo
- Sweden (11):
  - Södra Älvsborg Hospital, Borås
  - Eskilstuna Hospital, Eskilstuna
  - Sahlgrenska University Hospital, Gothenburg
  - Blekinge Hospital, Karlskrona
  - Skåne University Hospital, Lund
  - Örebro University Hospital, Örebro
  - Karolinska University Hospital, Stockholm
  - Sundsvall Hospital, Sundsvall
  - Umeå University Hospital, Umeå
  - Uppsala University Hospital, Uppsala
  - Central Hospital Växjö, Vaxjo

IPD SHARING:
Plan to Share IPD: No